CLINICAL TRIAL: NCT04658862
Title: A Phase 3, Multi-center, Randomized Study Evaluating Efficacy of TAR-200 in Combination With Cetrelimab Versus Concurrent Chemoradiotherapy in Participants With Muscle-Invasive Urothelial Carcinoma (MIBC) of the Bladder Who Are Not Receiving Radical Cystectomy
Brief Title: A Study of TAR-200 in Combination With Cetrelimab Versus Concurrent Chemoradiotherapy in Participants With Muscle-invasive Bladder Cancer (MIBC) of the Bladder
Acronym: SunRISe-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108917; 17000139BLC3001 (Other: Janssen Research & Development, LLC); 2020-002620-36 (EudraCT Number); 2023-507188-21-00 (Registry Identifier: EUCT number)
Expanded Access: NCT06877676 (Approved for marketing)
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAR-200 + Cetrelimab (Experimental): Participants will receive intravesical TAR-200 every 3 weeks (21 days indwelling) for first 18 weeks and thereafter from Week 24 every 12 weeks through study Year 3 in combination with intravenous (IV) Cetrelimab.
  Interventions: Biological: Cetrelimab; Drug: TAR-200
- Chemotherapy (cisplatin or gemcitabine) + Radiation Therapy (Active Comparator): Participants will receive chemotherapy based on investigator's choice from either cisplatin intravenously once weekly for 4 to 6 treatment weeks or gemcitabine intravenously twice weekly for 4 to 6 treatment weeks as Standard of Care (SOC) along with radiation therapy from either conventional radiotherapy (64 Gray [Gy], bladder only) for up to 6.5 treatment weeks or hypo-fractionated radiotherapy (55 Gy, bladder only) for up to 4 weeks.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Radiation: Conventional radiation therapy; Radiation: Hypo-fractioned radiation therapy

INTERVENTIONS:
Biological: Cetrelimab — Participants will receive intravenous Cetrelimab.
  Other Names: JNJ-63723283
  Arms: TAR-200 + Cetrelimab
Drug: TAR-200 — Participants will receive intravesical TAR-200.
  Other Names: JNJ-17000139
  Arms: TAR-200 + Cetrelimab
Drug: Cisplatin — Participants will receive cisplatin intravenously.
  Arms: Chemotherapy (cisplatin or gemcitabine) + Radiation Therapy
Drug: Gemcitabine — Participants will receive gemcitabine intravenously.
  Arms: Chemotherapy (cisplatin or gemcitabine) + Radiation Therapy
Radiation: Conventional radiation therapy — Participants will receive conventional radiation therapy for bladder (64 gy).
  Arms: Chemotherapy (cisplatin or gemcitabine) + Radiation Therapy
Radiation: Hypo-fractioned radiation therapy — Participants will receive hypo-fractioned radiation therapy for bladder (55 gy).
  Arms: Chemotherapy (cisplatin or gemcitabine) + Radiation Therapy

SUMMARY:
The purpose of study is to compare bladder intact-event free survival (BI-EFS) in participants receiving TAR-200 in combination with intravenous (IV) cetrelimab versus concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ineligible for or have elected not to undergo radical cystectomy
* All adverse events associated with any prior surgery and/or intravesical therapy must have resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade less than (<) 2 prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0, 1, or 2
* Thyroid function tests are within the normal range per investigator assessment (or stable on hormone supplementation). Investigators may consult an endocrinologist for participant eligibility assessment in the case of equivocal or marginal test results
* Adequate bone marrow, liver, and renal function: Bone marrow function (without the support of cytokines or erythropoiesis-stimulating agent in preceding two weeks): Absolute neutrophil count (ANC) greater than or equal to (>=) 1,500/cubic millimeters (mm^3); Platelet count >=80,000/mm^3; Hemoglobin >=9.0 grams per deciliter (g/dL); Liver function: (Total bilirubin less than or equal to (<=) 1.5 * upper limit of normal (ULN) or direct bilirubin <= ULN for participants with total bilirubin levels greater than (>)1.5*ULN (except participants with Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL), and Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to (<=) 2.5* institutional ULN); Renal function: Creatinine clearance >=30 mL/min using the Cockcroft-Gault formula. 24-hour creatinine clearance test will also be accepted for estimating renal function in situations where Cockcroft-Gault formula is not a good predictor of estimating adequate renal function

Exclusion Criteria:

* Must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder. Ta/T1/Carcinoma in situ (CIS) of the upper urinary tract (including renal pelvis and ureter) is allowable if treated with complete nephroureterectomy more than 24 months prior to initiating study
* Must not have diffuse CIS based on cystoscopy and biopsy. Diffuse, or multi-focal, CIS is defined as the presence of at least 4 distinct CIS lesions in the bladder at the time of the Screening re-TURBT
* Participants must not have evidence of cT4b, or N1-3, or M1 disease based on local radiology staging (chest, abdomen, and pelvis must be performed using Computed tomography [CT] or Magnetic resonance imaging [MRI]) within 42 days prior to randomization
* Presence of any bladder or urethral anatomic feature that, in the opinion of the investigator, may prevent the safe placement, indwelling use, or removal of TAR 200
* Evidence of bladder perforation during diagnostic cystoscopy. Participant is eligible if perforation has healed prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from Randomization to the First Bladder Intact Event-free Survival (BI-EFS) event | Up to 8 years
  Time from randomization to the first BI-EFS event includes histologically proven presence of muscle-invasive bladder cancer (MIBC), clinical evidence of nodal or metastatic disease (as assessed by RECIST 1.1 criteria), radical cystectomy (RC), or death due to any cause.

SECONDARY OUTCOMES:
Metastasis-free survival (MFS) | Up to 8 years
  MFS is measured from time from randomization to first radiologic (as assessed by RECIST 1.1 criteria) evidence of metastatic disease or death due to any cause.
Overall Survival (OS) | Up to 8 years
  OS is defined as time from randomization to death.
Overall Response Rate (ORR) | Up to 8 years
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR). CR is defined as Negative biopsy, and Computed tomography/Magnetic resonance imaging (CT/MRI) showing no evidence of locally advanced or metastatic disease. PR (down-staging) is defined as biopsy proven non-muscle invasive disease (Ta, T1, Tis) and CT/MRI showing no evidence of locally advanced or metastatic disease. Non-Response (NR) includes those not achieving a CR or PR. Those who do not undergo a biopsy will be considered Non-Evaluable (NE).
Number of Participants with Adverse Events (AEs) According to Common Terminology Criteria for Adverse Events (CTCAE) | Up to 8 years
  Number of Participants with AEs by Severity as assessed by CTCAE version 5 will be reported. Grade refers to the severity of the AE as follows: Grade 1- Mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2- Moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental Activities of Daily Living (ADL); Grade 3- Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self-care ADL; Grade 4- Life-threatening consequences, urgent intervention indicated; Grade 5- Death related to AE.
Number of Participants with AEs by Severity according to Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) | Up to 8 years
  NCI PRO-CTCAE is a patient-reported item library used to evaluate symptomatic treatment-emergent adverse events in participants on cancer clinical trials. The items selected for this study include all NCI PRO-CTCAE gastrointestinal items and urinary items. These items include taste changes, decreased appetite, nausea, vomiting, heartburn, gas, bloating, hiccups, constipation, diarrhea, abdominal pain, fecal incontinence, painful, urination, urinary urgency, urinary frequency, change in usual urine color, and urinary incontinence.
Number of Participants with Clinical Laboratory Abnormalities | Up to 8 years
  Number of participants with clinical laboratory abnormalities will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (290):
- United States (28):
  - Loma Linda Univ Faculty Medic, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Providence Saint John s Health Center, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology - Golden Off, Golden, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Urological Research Network, Hialeah, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - DuPage Medical Group, Lisle, Illinois
  - University Hospitals Seidman Cancer Center, Ann Arbor, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Adult Pediatric Urology & Urogynecology, P.C, Omaha, Nebraska
  - Garden State Urology, Morristown, New Jersey
  - New Jersey Urology LLC, Voorhees Township, New Jersey
  - Cardiology Clinic at Montefiore Hutchinson Complex, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vidant Urology - Greenville, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - University of Texas Medical Branch, League City, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (11):
  - Fundacion Intecnus, Bariloche
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Asociacion de Beneficencia Hospital Sirio Libanes, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Centro de Urologia (CDU), Ciudad Automoma Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Sanatorio Allende Cerro, Córdoba
  - Centro Oncologico Riojano Integral (Cori), La Rioja
  - Centro de Investigacion Pergamino SA, Pergamino
  - CEDIC Centro de Investigaciones Clinicas, Viedma
- Flinders Medical Centre, Bedford Park, Australia
- Austria (3):
  - Krankenhaus der barmherzigen Schwestern, Linz
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
  - Medizinische Universitaet Wien, Vienna
- Belgium (6):
  - Hopital Erasme, Anderlecht
  - ZNA Middelheim, Antwerp
  - AZ Sint-Lucas, Assebroek
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - Az Groeninge, Kortrijk
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (21):
  - Fundacao Pio XII, Barretos
  - Fundação Hospitalar São Francisco de Assis, Belo Horizonte
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Centro Regional Integrado de Oncologia CRIO, Fortaleza
  - Clinica de Oncologia Reichow, Jardim Blumenau
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital Regional do Cancer - Hospital de Esperança, Presidente Prudente
  - Hospital Sao Rafael, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Sociedade Beneficente de Senhoras - Hospital Sirio Libanes, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Centro Oncológico do Triângulo, Uberlândia
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec L Hotel Dieu de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- China (24):
  - Chinese Academy of Medical Sciences(CAMS) & Peking Union Medical College(PUMC), Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central Sourth University, Changsha
  - Hunan Cancer hospital, Changsha Shi
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Hospital of Jiaxing, Jiaxing
  - Nanjing Drum Tower Hospital, Nanjing
  - Qingdao Municipal Hospital, Qingdao
  - Ruijin Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Wuhan Tongji Hospital Tongji Medical College, Wuhan
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Czechia (8):
  - Slezska nemocnice v Opave, Opava
  - Fakultni nemocnice Plze, Plzen-Bory
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Urocentrum Praha, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Thomayerova nemocnice, Prague
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce, Prague
- France (22):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - ICH Hopital A. Morvan, Brest
  - Hôpital Côte de Nacre, Caen
  - Pole Sante Leonard de Vinci, Chambray-lès-Tours
  - Clinique Sainte Marguerite, Hyères
  - CHRU Lille, Lille
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Européen, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Tenon, Paris
  - Clinical La Croix Du Sud - Ramsay Santé, Quint-Fonsegrives
  - Centre hospitalier universitaire de St Etienne, Saint-Etienne
  - Centre Hospitalier Prive, Saint-Grégoire
  - Hopital Foch, Suresnes
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (15):
  - Klinikum Augsburg, Augsburg
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Urologicum Duisburg, Duisburg
  - Universitatsklinikum Dusseldorf, Düesseldorf
  - Klinik und Poliklinik für Urologie, Essen
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt am Main
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn - Klinikum am Gesundbrunnen, Heilbronn
  - Klinikum Herne - Urologie, Herne
  - Matthias Schulze - Germany, Markkleeberg
  - Universitatsklinikum Munster, Münster
  - Klinikum Nürnberg Nord - Hautklinik, Nuremberg
  - Krankenhaus der Barmherzigen Bruder Trier, Trier
- Greece (9):
  - Alexandra General Hospital of Athens, Athens
  - Metropolitan General A E, Cholargós
  - Athens Medical Center, Marousi
  - Metropolitan Hospital, Neo Faliro
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - Euromedica General Clinic, Thessaloniki
  - Clinic Agios Loukas, Thessaloniki
  - Papageorgiou General Hospital Of Thessaloniki, Thessaloniki
  - Anassa General Clinic, Volos
- Hungary (5):
  - Eszak Pesti Centrumkorhaz Honvedkorhaz, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
- India (9):
  - Sujan Surgical Cancer Hospital & Amravati Cancer Foundation, Amravati
  - Bangalore Medical College and Research Institute, Bangalore
  - Acharya Tulsi Regional Cancer Treatment Research Institute, Bikaner
  - Shatabdi Super Speciality Hospital, Nashik
  - BLK Super Specialty Hospital, New Delhi
  - Aakash Healthcare Super Speciality Hospital, New Delhi
  - Rajiv Gandhi Cancer Institute & Research Centre, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Jehangir Clinical Development Center Pvt Ltd, Pune
- Italy (24):
  - Ospedale San Donato, Arezzo
  - Fondazione del Piemonte per I Oncologia IRCC Candiolo, Candiolo
  - Ospedale Civile Ramazzini, Carpi
  - Ospedale Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - SPDC Villa Scassi, Genova
  - Ospedale San Martino, Genova
  - Ospedale Umberto I di Lugo, Lugo
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Sanitaria Locale Salerno - Po Andrea Tortora Di Pagani, Pagani
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - ASL Napoli 2 Nord-SM delle Grazie Hospital, Pozzuoli
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - Universita Campus Bio-Medico di Roma, Rome
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Istituto Clinico Humanitas Rozzano, IRCCS, Rozzano
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte, Siena
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale San Bortolo, Vicenza
- Japan (13):
  - Aso Co.,Ltd Iizuka Hospital, Iizuka
  - St Marianna University Hospital, Kanagawa
  - Nara Medical University Hospital, Kashihara
  - Saitama Medical University Hospital, Kawagoe-Shi
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Nagasaki University Hospital, Nagasaki
  - JOHAS Osaka Rosai Hospital, Osaka
  - Tokuyama Central Hospital, Shūnan
  - Toranomon Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Yamaguchi University Hospital, Ube
  - Yokohama City University Medical Center, Yokohama
- Mexico (11):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Consultorio Privado Dr Jose Arturo Rodriguez Rivera, Guadalajara
  - Centro De Estudio Y Prevencion Del Cancer, Juchitán de Zaragoza
  - Dr. Marco Antonio Badillo Santoyo, León
  - Oncologia Integral Satelite, Mexico City
  - i Can Oncology Center, Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Oncologico Potosino, San Luis Potosí City
  - Investigación Biomedica para el desarrollo de Farmacos, S.A. de C.V., Zapopan
- Poland (4):
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Siedlce
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar e Universitario de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Fund. Champalimaud, Lisbon
  - H. Santa Maria - Centro Hospitalar de Lisboa Norte, Lisbon
  - Hospital de Sao Joao, Porto
- Russia (12):
  - Altlay Regional Oncology Dispensary, Barnaul
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Krasnoyarsk Regional Oncology Dispensary, Krasnoyarsk
  - Hertzen Oncology Research Institute, Moscow
  - A. Tsyb Medical Radiological Research Center, Obninsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - Ryazan State Medical University named after I.P.Pavlov, Ryazan
  - N.N. Petrov Research Institute Of Oncology, Saint Petersburg
  - Ogarev Mordovian State University, Saransk
  - State Medical Institution Oncological Center #2 of Healthcare Department at Krasnodar Regio, Sochi
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - Bashkir State Medical University, Ufa
- South Korea (13):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Samsung Medical Center, Gangnam Gu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Namdong
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (14):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Fund. Puigvert, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Instituto Valenciano de Oncologia, Valencia
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (7):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Adana Baskent Yuregir Hospital, Adana
  - Yildirim Beyazit University Medical Faculty Ankara Atatürk Research and Training Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Dokuz Eylul Universitesi Tip Fakultesi, Balçova
  - Bezmialem University Medical Faculty, Fatih
  - Medical Park Gaziantep Hastanesi, Gaziantep
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul
  - Izmir Medical Park Hospital, Izmir
  - Inonu University Medical Faculty, Malatya
  - Erciyes Univ MKD Hospital, Melikgazi
  - T.C. Saglik Bakanligi Ankara Numune Egitim ve Arastirma Hastanesi, Seyhan
- Ukraine (9):
  - Chernihivskyi oblasnyi onkolohichnyi dyspanser, Chernihiv
  - SE Dnipropetrovsk Medical Academy, Dnipro
  - Kharkiv Regional Clinical Hospital, Kharkiv
  - Khersonsky Regional Oncology Center, Kherson
  - Asklepion LLC, Kiev
  - Kyiv City Clinical Hospital #3, Kyiv
  - State Institution Academy Of Medical Sciences Of Ukraine, Kyiv
  - P.L. Shupyk National Medical Academy of Post-Graduate Education, Kyiv
  - Lviv Regional Clinical Hospital, Lviv

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency